CLINICAL TRIAL: NCT06884852
Title: Ultrasound-guided Multilevel Erectorspinae Plane Block Versus Thoracic Epidural Analgesia for Prevention of Post Mastectomy Pain Syndrome for Breast Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Dr Ahmed elsayeh, Assistant Lecturer of Anesthesiology, Surgical Intensive Care Unit and Pain Medicine, National Cancer Institute ,Cairo University, Egypt, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AP2405-201-046-193
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Ultrasound; Multilevel Erector Spinae Plane Block; Thoracic Epidural Analgesia; Post Mastectomy; Pain Syndrome; Breast Cancer Patients
MeSH Terms: conditions — Somatoform Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block (ESPB) (Experimental): Erector spinae plane block (ESPB) using multilevel injections of bupivacaine 0.25%.
  We injected 15ml at the level of T2 and 15ml at the level of T5.
  Interventions: Drug: Erector spinae plane block (ESPB)
- Thoracic epidural block (Experimental): Thoracic epidural block at level of T5 -T6 using 10 ml of bupivacaine 0.25% as a bolus followed by 5 ml bupivacaine 0.25% every 1-2 hours depending on the duration of surgery and the response of the patient.
  Interventions: Drug: Thoracic epidural block

INTERVENTIONS:
Drug: Erector spinae plane block (ESPB) — Erector spinae plane block (ESPB) using multilevel injections of bupivacaine 0.25%.
  We will inject 15ml at the level of T2 and 15ml at the level of T5.
  Other Names: Bupivacaine 0.25%
  Arms: Erector spinae plane block (ESPB)
Drug: Thoracic epidural block — Thoracic epidural block at level of T5 -T6 using 10 ml of bupivacaine 0.25% as a bolus followed by 5 ml bupivacaine 0.25% every 1-2 hours depending on the duration of surgery and the response of the patient.
  Other Names: Bupivacaine 0.25%
  Arms: Thoracic epidural block

SUMMARY:
The aim of this study is to compare the analgesic efficacy of multilevel erector spinae plane block (ESPB) vs thoracic epidural in modified radical mastectomy (MRM) regarding duration of analgesia, postoperative opioid consumption, effect on intraoperative fentanyl consumption, postoperative numerical pain rating scale and quality of life for the next 6 months.

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy among females. Modified Radical Mastectomy (MRM) is the principal surgical treatment for breast cancer. The standard mode of anesthesia is general anesthesia, in addition to regional blocks for effective postoperative pain control.

Pain is usually managed by narcotics, which have many side effects, including prolonged sedation, increasing incidence of pain recurrence, respiratory depression, nausea & vomiting and paralytic ileus. All requiring close monitoring and in some occasions Intensive Care Unit (ICU) admission. Thoracic epidural and paravertebral blocks are the gold standard techniques. However, both techniques may lead to some serious complications including spinal cord injury, pneumothorax, incompatibility with pre-existing anticoagulation or antiplatelet therapy and hemodynamic instability.

Recently, multiple regional techniques have been used for postoperative thoracic pain control, including that caused by modified radical mastectomy. Interfascial plane blocks are currently the hot topic in management of postoperative pain. One of these blocks is erector spinae plane block (ESPB). It is an interfacial Para spinal plane block that is simple, safe, effective and associated with fewer complications in comparison to the gold standard techniques.

ELIGIBILITY:
Inclusion Criteria:

* Female patients age ≥ 18 years and ≤ 65 Years.
* Type of surgery; Modified Radical Mastectomy (MRM)
* Physical status ASA II, III.
* Body mass index (BMI): > 20 kg/m2 and < 35 kg/m2.

Exclusion Criteria:

* Patient refusal.
* Allergy or a contraindication to the drug used in the study, e.g. local anesthetics, opioids.
* History of psychological disorders.
* History of chronic pain.
* Contraindication to regional anesthesia e.g. sepsis, peripheral neuropathies and coagulopathy.
* Advanced chronic renal disease, which is defined as a chronic kidney disease (CKD) in which there is a severe reduction in glomerular filtration rate (GFR < 30 ml/min) and includes stages 4 and 5 of the CKD classification.
* Decompensated cirrhosis, which is defined as an acute deterioration in liver function in a patient with cirrhosis and is characterized by jaundice, ascites, hepatic encephalopathy, hepatorenal syndrome, or variceal hemorrhage.
* Severe heart disease which is defined as NYHA class iii (moderate symptoms with less than normal activity, marked limitation of function status) or NYHA class IV (severe symptoms with features of heart failure with minimal activity or at rest and severe limitation of functional status)
* Severe lung disease which includes oxygen saturation of blood less than 92%, RR more than 20, FEV1/FVC ratio less than 60%.
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients
Enrollment: 44 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
The average duration of analgesia | 24 hours postoperatively
  The average duration of analgesia will be recorded from the end of surgery till the first dose of morphine administrated.

SECONDARY OUTCOMES:
The total amount of morphine | 24 hours postoperatively
  Patient will be discharged to the ward then rescue analgesia will be given in the form of IV morphine 3 mg boluses if the patient reported Numeric Pain Rating Scale ≥ 4. The total amount of morphine given in 24 hours will be recorded for the two groups.
Incidence of postmastectomy pain syndrome | 6 months postoperatively
  Incidence of postmastectomy pain syndrome at 1, 3, and 6 months postoperatively will be recorded.
The total amount of fentanyl | Intraoperatively
  Fentanyl 1 μg/kg will be given if the mean arterial blood pressure or heart rate rises above 20% of the baseline levels.
Heart rate (HR) | 24 hours Postoperatively
  Heart rate will be noted at 4, 8, 12, 16, 20, and 24 hours postoperatively
Mean arterial blood pressure (MAP) | 24 hours Postoperatively
  Mean arterial blood pressure will be noted at 4, 8, 12, 16, 20, and 24 hours postoperatively
Degree of pain | 24 hours Postoperatively
  Each patient will be instructed about postoperative pain assessment with the numeric rating scale (NRS) score. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS will be recorded (at rest and during movement) at 0, 4, 8, 12, 16, 20, and 24 hours postoperatively.
Incidence of Postoperative nausea and vomiting (PONV). | 24 hours Postoperatively
  Postoperative nausea and vomiting (PONV) will be rated on a four-point verbal scale; (none =no nausea, mild = nausea but no vomiting, moderate= vomiting one attack, severe =vomiting > one attack). 0.1 mg/kg of IV ondansetron will be given to patients with moderate or severe postoperative nausea and vomiting.Nausea and vomiting Scores using a four-point verbal scale; on arrival to post-anesthesia care unit (PACU), scoring at 0, 4, 8,12,16,20 and 24 hours postoperatively.
Complications related to the block | 6 months postoperatively
  Complications related to the block such as local anesthetics, systemic toxicity, and vascular injury will be recorded
Morphine-related complications | 24 hours Postoperatively
  Patient will be discharged to the ward then rescue analgesia will be given in the form of IV morphine 3 mg boluses if the patient reported Numeric Pain Rating Scale ≥ 4. The total amount of morphine given in 24 hours will be recorded for the two groups. Morphine-related complications such as respiratory depression, urine retention, or pruritis will be recorded.
Patient's satisfaction | 24 hours Postoperatively
  Patient's satisfaction: the patient will be classified in this group as satisfied or not.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author